CLINICAL TRIAL: NCT02273687
Title: Analysis of Time-motion-mode Ultrasound Diaphragm Measures in Patients With Acute Respiratory Distress in Emergency Department: Predicting Respiratory Prognosis
Brief Title: Time-motion-mode Ultrasound Diaphragm Measures in Patients With Acute Respiratory Distress in Emergency Department
Acronym: EDDRAPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/20143/XBAC-01; 2014-A00511-46 (Other: ANSM)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: diaphragm movement; ultrasound; emergency room
MeSH Terms: conditions — Respiratory Distress Syndrome; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prognostic study population (Experimental): The study population consists of patients treated for acute respiratory distress in the emergency department at the Nîmes University Hospital. See inclusion and exclusion criteria.
  Intervention: Diaphragmatic ultrasound
  Interventions: Device: Vivid S6 GE Ultrasound

INTERVENTIONS:
Device: Vivid S6 GE Ultrasound — Diaphragmatic ultrasound will be performed by the physician supporting the patient on arrival and also at 4 hours later in the beginning of therapeutic management. The patient will be monitored for 24 hours following inclusion.
  The exams will all be done with the same ultrasound system (Vivid S6 GE Ultrasound) and a phased array probe, also called a cardiac probe.

SUMMARY:
The main objective of this study is to show that "diaphragmatic excursion measures upon emergency admission" (CDA values) on patients with acute respiratory failure are predictive of the need to use mechanical ventilation (invasive or non-) in the first four hours.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A-determine a prognostic threshold for diaphragmatic excursion measures able to predict the use of mechanical ventilation (invasive or not) in the first four hours.

B-to study the association between CDA values and persistence of respiratory distress during the first 4 hours of care among patients who, at 4 hours, are not mechanically ventilated.

C-to study the association between CDA values and respiratory re-exacerbation or a continuing need for mechanical ventilation during the 24 first hours after admission to the emergency room D-to study the association between diaphragmatic excursion measures made after initial emergency care (at 4 hours; =CDH4), and the persistence of respiratory distress at 4 hours, in patients who at 4 hours are not mechanically ventilated.

E-to study the association between CDH4 values and respiratory re-exacerbation during the 24 first hours after admission to the emergency room among patients who, at 4 hours, are not mechanically ventilated F-to study the association between changes in values of diaphragmatic excursion measure before and after initial emergency care (CDA → CDH4) and respiratory re-exacerbation during the 24 first hours after admission to the emergency room among patients who, at 4 hours, are not mechanically ventilated.

G-analyze patient outcomes by subgroup according to diagnosis (decompensated COPD, OAP, lung disease, asthma, pleural disease).

ELIGIBILITY:
Inclusion Criteria:

* The patient has given informed consent (and signed the consent form) or, in case of an emergency situation, an investigator has committed to obtaining the consent of the patient as soon as his/her condition permits
* Patient affiliated with or beneficiary of a health insurance plan
* Acute Respiratory Distress (DRA) defined by: (1) respiratory rate > 25 and/or signs of struggle and hypoxia AND (2) SpO2 values < 90% and/or [pH < 7.35 and pCO2 > 6 kPa (45 mm Hg)]
* Breathing spontaneously (no ventilation)

Exclusion Criteria:

* Patient currently participating in or having participated in another interventional study in the previous three months, or patient in an exclusion period determined by a previous study
* Patient under judicial protection or any kind of guardianship
* Refusal to sign the consent
* Patient pregnant, parturient, or lactating
* Neurological or neuromuscular disease modifying the operation of the diaphragm without any decompensation (Polyneuropathy, Lou Gehrig's disease, Myasthenia ...)
* Patient who received mechanical ventilation at home
* Patient who received treatment by mechanical ventilation during the pre-hospitalization care phase
* Patient admitted with respiratory failure requiring immediate installation of a mechanical ventilation and thus not allowing the performance of two ultrasound measurements
* Patient suffering from a pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Measurement of diaphragmatic excursion by M-mode ultrasound | Day 0, baseline
  in centimeters
Use of ventilation within the first 4 hours | Day 0, baseline + 4 hours
  yes/no

SECONDARY OUTCOMES:
Measurement of diaphragmatic excursion by M-mode ultrasound | Day 0, baseline + 4 hours
  in centimeters
Acute respiratory distress signs within the first 4 hours | Day 0, baseline + 4 hours
  yes/no
Signs of respiratory re aggravation at 24 hours | Day 1
  yes/no
Diagnosis | Day 1
  qualitative variable: decompensated COPD, OAP, pneumonia, asthma, or pleural pathology

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CH de Perpignan - Hôpital Saint Jean, Perpignan

REFERENCES:
- [Result] Clement A, Zieleskiewicz L, Bonnec JM, Occean BV, Bastide S, Muller L, de La Coussaye JE, Boussuges A, Claret PG, Bobbia X. Diaphragmatic excursion measurement in emergency department patients with acute dyspnea to predict mechanical ventilation use. Am J Emerg Med. 2020 Oct;38(10):2081-2087. doi: 10.1016/j.ajem.2020.06.044. Epub 2020 Jun 26. PMID 33142179